CLINICAL TRIAL: NCT05953961
Title: Randomized Study of Therapshere 90-Yittrium Transarterial Radioembolization Versus Microwave Ablation in Small Hepatocellular Carcinoma With Hypoalbuminemia
Brief Title: 90Y Transarterial Radioembolization Versus Microwave Ablation in Small Hepatocellular Carcinoma With Hypoalbuminemia
Acronym: REALM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.090; Sponsored Research Agreement (Other Grant/Funding Number: Boston Scientific)
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Yttrium-90; Hypoalbuminemia
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypoalbuminemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Therasphere Transarterial Radioembolization (Active Comparator): Two-phase treatment including mapping angiogram with personalized dosimetry followed by complete treatment of the tumor angiosome with 90-Yittrium glass microsphere infusion.
  Interventions: Device: Therasphere 90Y
- Microwave Ablation (Active Comparator): Ablation performed with a high powered, gas cooled multi-antenna system targeting an ablative margin > 5mm.
  Interventions: Device: Microwave Ablation

INTERVENTIONS:
Device: Therasphere 90Y — Transarterial Radioembolization
  Arms: Therasphere Transarterial Radioembolization
Device: Microwave Ablation — Microwave Ablation
  Arms: Microwave Ablation

SUMMARY:
This clinical trial will compare 1-year outcomes in patients with hypoalbuminemia and a new diagnosis of small, early-stage hepatocellular carcinoma (HCC) who are candidates for both 90-Yittrium Therasphere transarterial radioembolization (90Y) and microwave ablation (MWA). The study will determine whether treatment with 90Y lowers the risk of disease progression within the first year after diagnosis. Participants will be randomized to receive either first cycle 90Y or MWA and then proceed with standard of care.

DETAILED DESCRIPTION:
This study will compare 1-year outcomes in patients with hypoalbuminemia and a new diagnosis of early-stage hepatocellular carcinoma (HCC) who are candidates for both 90-Yittrium Therasphere transarterial radioembolization (90Y) and microwave ablation (MWA). The study will focus on patients with solitary, small HCC, defined as a single tumor ≤ 3cm in diameter, and with hypoalbuminemia at the time of HCC diagnosis, defined as albumin < 3.4 g/dL. Participants will be randomized to receive either 90Y or MWA as a first cycle liver-directed therapy.

The study will enroll 50 participants randomized at a 1:1 ratio to 90Y or MWA. After first cycle treatment, the participants will resume standard of care management for early-stage HCC. Participants will undergo observational follow-up for 1-year after first cycle treatment to collect data on adverse events, response to treatment, time to retreatment, duration of response, and progression of disease staging.

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosis according to the Liver Imaging - Reporting Data System (LI-RADS) Criteria as defined in the American Association for the Study of Liver Diseases 2018 HCC practice guidelines
* Eastern Cooperative Oncology Group score 0 - 1
* Child-Pugh A - B
* Bilirubin < 2.5 mg/dL
* Creatinine < 2.0 mg/dL
* No prior liver-directed therapy or systemic therapy for HCC
* Solitary, unresectable HCC ≤ 3cm
* Albumin level < 3.4 g/dL at HCC diagnosis
* Tumor anatomical location and angiosome amendable to MWA and 90Y

Exclusion Criteria:

* Pregnant women
* Concurrent malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Disease Progression | 1-year
  Progression in disease staging according to the Barcelona Clinic Liver Cancer Staging Algorithm

SECONDARY OUTCOMES:
Target Response Evaluation Criteria in Solid Tumors modified for HCC | 60 - 120 days post-treatment
  Durable target tumor response rate
Time to Retreatment | 1 year
  Duration of time following the first cycle treatment until the targeted tumor requires additional treatment
Duration of Response | 1 year
  Duration of time after first cycle treatment the target tumor continues to respond to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ari Cohen, MD, Principal Investigator — Ochsner Health
Locations (1):
- Ochsner Main Campus, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No